CLINICAL TRIAL: NCT06925516
Title: Efficacy and Safety of Apatinib Combined With Adebrelimab and GEMOX Regimen Chemotherapy as the First-line Treatment for Unresectable Intrahepatic Cholangiocarcinoma (ICC): A Single-arm, Multicenter, Phase II Study
Brief Title: A Trial of Apatinib and Adebrelimab in Combination With Chemotherapy in Patients With Unresectable ICC
Acronym: ACADEMY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-012-02
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc)
Keywords: unresectable intrahepatic cholangiocarcinoma; cholangiocarcinoma; GEMOX chemotherapy; Antineoplastic Agents; Tyrosine kinase inhibitors
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — apatinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib and Adebrelimab in Combination With chemotherapy (Experimental): Adebrelimab (IV 1200mg q3w) and apatinib (PO 250mg qd) plus GEMOX (up to 6 cycles) in 21day cycles
  Interventions: Drug: Apatinib and Adebrelimab in Combination With chemotherapy

INTERVENTIONS:
Drug: Apatinib and Adebrelimab in Combination With chemotherapy — Patients would receive Adebrelimab (IV 1200mg q3w) and apatinib (PO 250mg qd) plus GEMOX (up to 6 cycles) in 21day cycles. Apatinib and Adebrelimab would be maintained until the disease progressed or intolerable toxicity and adverse reactions or the medication was used for two years.

SUMMARY:
The study aims to evaluate the efficacy and safety of Apatinib and Adebrelimab in Combination With chemotherapy in patients with advanced intrahepatic cholangiocarcinoma (ICC)

DETAILED DESCRIPTION:
The investigators are conducting a clinical research study to evaluate the effectiveness and safety of a novel combination therapy for patients with advanced, unresectable intrahepatic cholangiocarcinoma (ICC). The study hypothesizes that combining three treatments, apatinib (an oral TKI selectively targeting VEGFR2) and adebrelimab (an immune checkpoint inhibitor) plus GEMOX chemotherapy (a standard chemotherapy regimen of gemcitabine and oxaliplatin), will significantly improve outcomes compared to traditional chemotherapy alone. The primary goal is to measure how many patients experience tumor response (objective response rate, ORR), with historical data suggesting a 16% response rate for chemotherapy alone, while this study aims to achieve a 40% response rate. Secondary goals include assessing how long patients live without cancer worsening (progression-free survival), overall survival, and monitoring side effects. The trial will enroll 38 participants across multiple hospitals, all of whom will receive the combination therapy for up to two years or until the cancer progresses or side effects become unmanageable. Researchers will also explore whether specific biological markers, such as tumor protein levels or genetic changes, predict better responses to the treatment. By testing this three-drug combination, the study seeks to provide a more effective and tolerable first-line option for a cancer type with limited treatment choices and poor survival rates.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provided informed consent and sign the informed consent form;
* 2. Male or female, Aged 18-75 years (counted on the date of signing informed consent);
* 3. Histologically or cytologically confirmed ICC;
* 4. The patient is not a candidate for surgery, or the disease has progressed after prior surgery and/or local treatment.
* 5. No previous systematic treatment for advanced ICC. Exceptions include patients who relapsed more than 6 months after adjuvant chemotherapy following radical resection. Local regional therapy (including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic arterial infusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection) must have been completed at least 4 weeks prior to baseline radiological scanning, and any toxicity (except alopecia) induced by local regional therapy must have resolved to ≤ Grade 1 in accordance with National Cancer Institute - Common Terminology Criteria for Adverse Event version 5.0 (NCI-CTCAE v5.0);
* 6. Have at least one measurable lesion (in accordance with RECIST v1.1, major diameter ≥ 10 mm of the measurable lesion in spiral CT scan or short diameter of swollen lymph node ≥ 15 mm; the lesion with previous local therapy can be used as target lesion after the progression is confirmed in accordance with RECIST v1.1)
* 7. Child-Pugh class: Grade A;
* 8. ECOG-PS score: 0-1;
* 9. With a life expectancy of ≥ 12 weeks;
* 10. Adequate major organ function without severe hematologic, cardiac, pulmonary, hepatic, renal, or bone marrow dysfunction, and no immunodeficiency disease;
* 11. If subjects have active hepatitis B (HBV) infection: HBV- deoxyribonucleic acid (DNA) must be < 500 IU/mL (or must be < 2500 copy/mL if copy/mL is the only unit available in the study site) and are willing to receive antiviral therapy throughout the study (treatment in accordance with local standard of care, e.g., entecavir);
* 12. Women of childbearing potential must agree to abstain from heterosexual intercourse or use reliable contraception from the time of signing informed consent until at least 120 days after the last study drug administration. A negative serum pregnancy test (HCG) must be confirmed within 7 days before starting study treatment. Lactating women are excluded;
* 13. Men with female partners of childbearing potential must agree to abstain from heterosexual intercourse or use reliable contraception from the time of signing informed consent until at least 120 days after the last study drug administration. Men must also agree not to donate sperm during this period. For men whose partners are pregnant, condom use is required without additional contraception;

Exclusion Criteria:

* 1. Known hepatocellular carcinoma, Combined Hepatocellular and Intrahepatic Cholangiocarcinoma, sarcomatoid hepatocellular carcinoma, fibrolamellar carcinoma of liver;
* 2. Other active malignant tumor except ICC within 5 years or simultaneously. Cured localized tumor, for example, basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of prostate, carcinoma in situs of cervix, breast cancer in situ may be enrolled;
* 3. Planning to or previously received organ or allogenic bone marrow transplantation;
* 4. Treatment of other investigational product(s) within 28 days prior to the start of study treatment;
* 5. Previous treatment with Immune Checkpoint Inhibitors: Prior use of any antibody/drug targeting T-cell co-regulatory proteins (immune checkpoints), including anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies (including topical use).
* 6. Moderate-to-severe ascites with clinical symptoms, i.e., requiring therapeutic puncture or drainage, or Child-Pugh score >2, except the subjects with small amount of ascites in radiological examination but free from clinical symptoms; uncontrolled or moderate to severe pleural effusion, pericardial effusion.
* 7. History of gastrointestinal bleeding within 6 months prior to the start of study treatment or clear tendency of gastrointestinal bleeding;
* 8. Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment;
* 9. Known genetic or acquired hemorrhage (e.g., coagulation dysfunction) or thrombotic tendency, for example, subject with hemophilia; current or recent (within 10 days prior to the start of study treatment) use of full-dose of oral or intravenous anticoagulant or thrombolytic drug for the purpose of treatment (preventive use of low-dose aspirin or low molecular weight heparin is allowed);
* 10. Current or recent (within 10 days prior to the start of study treatment) use of aspirin (> 325 mg/day, maximum dose for antiplatelet) or dipyridamole, ticlopidine, clopidogrel and cilostazol;
* 11. Thrombosis or thromboembolic event within 6 months prior to the start of study treatment, for example, cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism;
* 12. Cardiac clinical symptom or disease that is not well controlled;
* 13. Hypertension that cannot be well controlled through antihypertensive drugs, allowing to reach the above parameters by the use of antihypertensive therapy; previous hypertensive crisis or hypertensive encephalopathy;
* 14. Major vascular disease within 6 months prior to the start of study treatment (for example, aortic aneurysm requiring surgical repair or peripheral arterial thrombosis in recent days); Serious, unhealed or splitting wound and active ulcer or untreated bone fracture; Major surgical therapy within 4 weeks prior to the start of study treatment (except diagnosis), or planned major surgery during the study;
* 15. Evidence on intraperitoneal pneumatosis that can not be explained by puncture or recent surgery;
* 16. Previous or current presence of metastasis to central nervous system; Metastatic disease involving main airway or blood vessels (e.g. Vena cava tumor invasion or complete occlusion of the major portal vein due to HCC, the major portal vein is defined as the part of portal vein between the union of the splenic and superior mesenteric veins and the first bifurcation into the left and right vein) or high-volume mediastinal tumor mass located in the center (distance from carina <30 mm);
* 17. History of hepatic encephalopathy; Current interstitial pneumonia or interstitial lung disease, or history of interstitial pneumonia or interstitial lung disease which required hormonal therapy, or other pulmonary fibrosis that may interfere with the judgement and treatment of immune-related pulmonary toxicity; organizing pneumonia (e.g., obliterative bronchiolitis), pneumoconiosis, drug related pneumonitis, idiopathic pneumonia, subjects with evidence on active pneumonia or serious pulmonary function impairment on thoracic computed tomography (CT) in screening period (previous radiation pneumonitis in the radiation area will be allowed); active tuberculosis;
* 18. Active autoimmune disease or history of autoimmune disease and may relapse (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [with the exception that it can be controlled by hormone replacement therapy]). Subjects with skin disease that do not require systemic treatment are eligible, for example, leukoderma, psoriasis, alopecia; subjects with controlled type 1 diabetes by insulin are eligible; subjects with asthma that has been completely resolved in childhood and don't need any treatment are eligible, but subjects with asthma that require a bronchodilator as medical intervention are not eligible;
* 19. Use of immunosuppressive medication within 14 days prior to the start of study treatment, or systemic corticosteroid therapy to achieve the objective of immunosuppression (Prednisone at the dose of >10mg/day or equivalent);
* 20. Known history of hypersensitivity to the active substance or to any other components of each investigational medicinal product;
* 21. Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteremia or complications of severe pneumonia; oral or intravenous therapeutic antibiotics within 2 weeks prior to the start of study treatment (subjects who are treated with antibiotics for prevention, e.g., preventive urinary tract infection or exacerbation of chronic obstructive pulmonary disease are eligible for participation in the study);
* 22. Congenital or acquired immunodeficiency (e.g., HIV infection);
* 23. Hepatitis B and hepatitis C co-infection;
* 24. Attenuated live vaccine therapy administered within 28 days prior to the start of study treatment, or are expected to receive such vaccines during Adebrelimab treatment or within 60 days after the last dose of Adebrelimab;
* 25. Other factors that may affect the study results or lead to early study termination as judged by investigators, such as alcoholism, drug abuse, other serious diseases (including mental disorders) requiring concomitant therapy, with serious laboratory examination abnormality, with family or social factors, that may affect subject's safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 12 months
  the objective response rate (ORR) of advanced ICC patients who progressed after standard treatment with Adebrelimab and apatinib plus GEMOX.

SECONDARY OUTCOMES:
Adverse Events | from the first drug administration to within 30 days for the last Adebrelimab dose
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v5.0
progression free survival (PFS) | up to 24 months
  PFS was defined as the time from the start of treatment to the date of first documentation of disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST v1.1), or date of death, whichever occurred first.
overall survival (OS) | up to 24 months
  OS is the time interval from the start of treatment to death due to any reason or loss of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Changzhen Shang, M.D, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No